CLINICAL TRIAL: NCT05916820
Title: Effects of Tanzberger Versus Pelvic Floor Muscle Training on Urinary Incontinence and Quality of Life in post_menopausal Females
Brief Title: Effects of Tanzberger Versus Pelvic Floor Muscle Exercises on Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Iqra Shafi
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Urinary Incontinence; Menopause
Keywords: Pelvic floor muscle training; Tanzberger Exercise; Urine Incontinence
MeSH Terms: conditions — Urinary Incontinence; Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tanzberger Exercises (Experimental): It consist of patients who will receive Tanzberger exercises 3 sessions per week for 4 weeks.
  Interventions: Other: Tanzberger Exercises
- Pelvic floor muscle training (Experimental): It consists of patients who will receive pelvic floor muscle training 3 sessions per week for 4 weeks.
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Other: Tanzberger Exercises — It consists of patients who will receive Tanzberger exercise 3 sessions per week for 4 weeks. e.g. Rolling on the ball forward, Back to back sitting.
  Arms: Tanzberger Exercises
Other: Pelvic floor muscle training — It consists of patients who will pelvic floor muscles exercise 3 sessions per week for 4 weeks. e.g. Assisted heel drop, Bridge, Dead Bug, Bird DOG
  Arms: Pelvic floor muscle training

SUMMARY:
Randomized clinical trial (RCT) will be conducted to compare the effects of Tanzberger exercises and pelvic floor muscle training on urinary incontinence and quality of life in post_menopausal females suffering from urine incontinence in which data will be collected from Razahat Medical Centre, Lahore via International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form score (ICIQ-UI-SF) and incontinence quality of life (IQOL) Questionnaire. Sample size of 34 patients will be taken. Non_probability convenient sampling will be used. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups through lottery method, to either the PFMs group or Tanzberger exercise group. Treatment will be given three times a week. International Consultation on Incontinence Questionnaire, Urinary Incontinence-Short Form Questionnaire and Incontinence quality of life will be used to measure quality of life. All participants in both groups will be evaluated before and after the treatment programs. Total duration of study will be six months. Data will be analyzed by using SPSS 21

DETAILED DESCRIPTION:
Urinary Incontinence is defined by the International Continence Society (ICS) as the involuntary loss of urine through urethra which is distressing and disabling condition mainly affecting the social and psychological well-being of an individual. Due to the embarrassing nature of incontinence, it is both underreported and under diagnosed. It affects women's quality of life. Tanzberger technique using Swiss ball strengthen levator ani muscles which play role in closing urethra. Pelvic floor muscle exercises are safe and efficient treatment option to treat urinary incontinence and improves quality of life. The significance of this study is, PMFs training and Tanzberger exercises will be executed in comparison to treat post-menopausal women who are facing with unhygienic and social embarrassing health disorder of Urinary Incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 to 60 years.
* Postmenopausal Females
* Diagnosed patients of urinary incontinence

Exclusion Criteria:

* Delivery with any complication.
* Females have any history of diabetes, hypertension, neurological, or any chronic illness.
* Any pelvic or abdominal surgery
* Disc herniation or spine fracture.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Incontinence Quality of life questionnaire | 4th week
  The I-QoL Questionnaire consists of 22 questions that assess the limitations on human behavior, the psychosocial impact and social constraint brought about by urinary incontinence. Responses are given on a scale ranging from 1 to 5 points and the final scores are then summed up and converted into percentages. The higher the percentage, the better the quality of life. Reliability was assessed by Cronbach's alpha(0.93)
International Consultation on Incontinence Questionnaire-Urinary Incontinence | 4th week
  The ICIQ-UI-SF measures the degree of urinary incontinence and gives it a score on a range of 0 - 21, where higher numbers in any part indicate a worse urinary incontinence. This questionnaire examines the frequency, amount and duration of urine leakage and its effect on the quality of life. Numerous studies used this tool and its reliability and validity were confirmed in Iran with a Cronbach's alpha of 0.75

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, MS, Principal Investigator — Riphah International University
Locations (1):
- Razahat Medical Center,Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez Isaza P, Jaguszewska K, Cardona JL, Lukaszuk M. Long-term effect of thermoablative fractional CO2 laser treatment as a novel approach to urinary incontinence management in women with genitourinary syndrome of menopause. Int Urogynecol J. 2018 Feb;29(2):211-215. doi: 10.1007/s00192-017-3352-1. Epub 2017 May 18. PMID 28523400
- [Background] Vaughan CP, Markland AD. Urinary Incontinence in Women. Ann Intern Med. 2020 Feb 4;172(3):ITC17-ITC32. doi: 10.7326/AITC202002040. PMID 32016335
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322